CLINICAL TRIAL: NCT01224015
Title: Safety and Efficacy Study of Botulinum Toxin Type A for the Treatment of Crow's Feet Lines and Frown Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-104; 2010-021271-83 (EudraCT Number)
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Facial Rhytides; Crow's Feet Lines; Glabellar Lines
MeSH Terms: interventions — Saline Solution; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- onabotulinumtoxinA 24U (Other): 24 units (U) onabotulinumtoxinA (botulinum toxin Type A) total dose and placebo injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients may receive up to 2 treatments during the study.
  Interventions: Drug: normal saline; Biological: onabotulinumtoxinA 24 U
- placebo (normal saline) (Placebo Comparator): Normal Saline (placebo) injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients may receive up to 2 treatments during the study.
  Interventions: Drug: normal saline
- onabotulinumtoxinA 44U (Experimental): 44 units onabotulinumtoxinA (botulinum toxin Type A) total dose injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients may receive up to 2 treatments during the study.
  Interventions: Biological: onabotulinumtoxinA 44 U

INTERVENTIONS:
Drug: normal saline — Normal Saline injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients may receive up to 2 treatments during the study.
  Arms: onabotulinumtoxinA 24U; placebo (normal saline)
Biological: onabotulinumtoxinA 44 U — 44 units onabotulinumtoxinA (botulinum toxin type A) total dose injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients may receive up to 2 treatments during the study.
  Other Names: BOTOX®; BOTOX® Cosmetic; onabotulinumtoxinA
  Arms: onabotulinumtoxinA 44U
Biological: onabotulinumtoxinA 24 U — 24 units onabotulinumtoxinA (botulinum toxin type A) total dose injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients may receive up to 2 treatments during the study.
  Other Names: BOTOX®; BOTOX® Cosmetic; onabotulinumtoxinA
  Arms: onabotulinumtoxinA 24U

SUMMARY:
This study will evaluate the safety and efficacy of botulinum toxin type A compared to placebo for the treatment of Crow's Feet Lines and Frown Lines (Facial Rhytides) for patients who successfully completed Study 191622-099.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed Study 191622-099

Exclusion Criteria:

* Known immunization or hypersensitivity to botulinum toxin of any serotype
* Anticipated need for treatment with botulinum toxin of any serotype during the study (except for study treatment)
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis
* Anticipated need for surgery or hospitalization during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Newport Beach, California, United States
- Vancouver, British Columbia, Canada
- Antibes, France
- Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Extension study for patients who participated in study 191622-099
Groups:
- onabotulinumtoxinA 44U: 44 units (U) onabotulinumtoxinA (botulinum toxin Type A) total dose injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients received up to 2 treatments during the study.
- onabotulinumtoxinA 24U: 24 units onabotulinumtoxinA (botulinum toxin Type A) total dose and placebo injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients received up to 2 treatments during the study.
- Placebo (Normal Saline): Normal Saline injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients received up to 2 treatments during the study.
Period: Overall Study
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Started | 361 | 227 | 96
Completed | 347 | 211 | 83
Not Completed | 14 | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 361 | 227 | 96 | 684
Age, Customized [Number; unit: Participants]
  <45 Years | 105 | 68 | 33 | 206
  45 to 65 Years | 241 | 148 | 59 | 448
  >65 Years | 15 | 11 | 4 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315 | 203 | 80 | 598
  Male | 46 | 24 | 16 | 86

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Grade of None or Mild at Maximum Smile Based on the Investigator Facial Wrinkle Scale Assessment of the Severity of Crow's Feet Lines
Description: The investigator assessed the severity of the patient's Crow's Feet Lines at maximum smile using the 4-point Facial Wrinkle Scale: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a score of none or mild at Day 30 is reported.
Time Frame: Day 30
Population: Participants from the Intent-to-treat population, consisting of all randomized participants with data available for analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Number analyzed (Participants) | 349 | 223 | 95
Percentage of participants | 63.6 | 56.5 | 1.1

ADVERSE EVENTS:
Description: The safety population (all randomized participants who received study drug) was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 6/349 | 1/223 | 1/95
Other Adverse Events (participants affected / at risk) | 44/349 | 23/223 | 15/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | onabotulinumtoxinA 44U (N=349) | onabotulinumtoxinA 24U (N=223) | Placebo (Normal Saline) (N=95)
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Infected bites (Infections and infestations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | onabotulinumtoxinA 44U (N=349) | onabotulinumtoxinA 24U (N=223) | Placebo (Normal Saline) (N=95)
Injection site haematoma (General disorders) | 20 | 11 | 6
Nasopharyngitis (Infections and infestations) | 6 | 9 | 6
Headache (Nervous system disorders) | 18 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.